CLINICAL TRIAL: NCT03146559
Title: Using EMG of the Healthy Hand to Control TENS of the Affected Hand in Hemiparetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nachum Soroker, MD (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Sponsor-Investigator, Nachum Soroker, MD, head, Department of neurologic rehabilitation, Loewenstein, Loewenstein Hospital
Organization: Loewenstein Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: loe003516CTIL
Record Dates: First submitted 2017-05-07; First posted 2017-05-10 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Stroke
Keywords: Cross education; EMG
MeSH Terms: conditions — Stroke | interventions — Electromyography; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMG and TENS (Experimental): Wireless Bluetooth EMG ("Myo") bracelet will be placed on the healthy forearm. A voluntary dorsi flexion of the healthy wrist produces data that will be transmitted to a PC and will be used to activate (via Arduino controller) a Transcutaneous Electric Nerve Stimulator (TENS), placed on the paretic forearm, that will stimulate wrist dorsi flexors.
  5 days per week, for 3 weeks, 15 minutes per day.
  Interventions: Device: EMG and TENS
- TENS only (Active Comparator): Custom-built software & hardware: PC + Arduino controller and Transcutaneous Electric Nerve Stimulator (TENS) device, will be used to stimulate wrist dorsi flexors of the paretic forearm.
  5 days per week, for 3 weeks, 15 minutes per day.
  Interventions: Device: TENS only

INTERVENTIONS:
Device: EMG and TENS — Healthy hand EMG signal measured while making voluntarily wrist dorsi flexion will activate TENS, which will be placed on the paretic forearm and will produce wrist dorsi flexion.
  Arms: EMG and TENS
Device: TENS only — Automatic TENS stimuli to the paretic dorsi flexors (i.e., producing wrist dorsi flexion).
  Arms: TENS only

SUMMARY:
The purpose of this study is to investigate learning transfer from the healthy hand to the paretic hand in stroke patients. EMG signals from the healthy hand - while performing wrist dorsi flexion movement - will be used to activate electric muscles stimulation of the dorsi flexors of the paretic hand.

DETAILED DESCRIPTION:
14 post-stroke subjects will be recruited from neurological rehabilitation department at Loewenstein rehabilitation hospital, Ra'anana, Israel. The patients will be randomly assigned to one of two groups: 1) Experimental group. 2) Control group. The 3 weeks intervention (15 sessions) in each group will include electric muscles stimuli (pulse rate 35-100Hz pulse width 200 microseconds, 5 sec on and 10 sec rest ) of the hemiparetic hand for 15 minutes. The patients in the experimental group will wear a wireless Bluetooth EMG ("Myo" bracelet) on their healthy forearm and when they will execute wrist dorsi flexion, the data will be transmitted to a PC which will be used to activate (via Arduino controller) a Transcutaneous Electric Nerve Stimulator (TENS) that is attached to the paretic dorsi flexors (electrodes are placed on the paretic forearm). The control group will get only automatic stimuli on the paretic forearm via the TENS.

The assessments will be done before the intervention, at the end of three weeks of intervention, and after 1 month from the end of the intervention (follow up).

The outcomes will include: active range of motion of fingers and wrist dorsi flexion (using cybermin 5DT glove for digital measures), upper limb section of Fugl-Meyer test, Box and Blocks test and Jebsen Taylor Hand Function Test. Only before the beginning of the intervention the sensory ability of the patient will be assessed using the Sensory section of Fugl-Meyer (FM) and Semmes-Weinstein filaments for superficial sensation. Normalized lesion data will be computed using the ABLE module within MEDx software (Medical Numerics).

Differences between groups will be calculated using t-tests or Mann-Whitney, depending on distribution of normality with corrections for multiple comparisons.

ELIGIBILITY:
Inclusion Criteria:

* First stroke
* Age 25-80 years
* Able to understand research instructions

Exclusion Criteria:

* Unstable clinical/metabolic state

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2017-05-25 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Change in active range of motion of wrist dorsi flexion and fingers extension | Baseline, after 3 weeks of intervention and one month after the end of the intervention (follow up).
  The ability of the paretic hand to produce active range of motion (ROM) of paretic fingers and wrist by using digital measurements with 5DT Cybermin glove.

SECONDARY OUTCOMES:
Change in Fugl-Meyer Assessment | Baseline, after 3 weeks of intervention and one month after the end of the intervention (follow up).
  Score of 66 point indicate normal motor functioning of upper limb
Change in Box and Blocks test | Baseline, after 3 weeks of intervention and one month after the end of the intervention (follow up).
  Number of cubes transferred from one side of cube (chamber) to the other side of the cube within a minute
Change in Jebsen Taylor Hand Function Test | Baseline, after 3 weeks of intervention and one month after the end of the intervention (follow up).
  Time of performance of different task, mimicking activity of daily living, is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Sivi Frenkel-Toledo, PhD, Study Director — Loewenstein Hospital
Locations (1):
- Loewenstain hospital, Raanana, Israel